CLINICAL TRIAL: NCT04066218
Title: Assessing Patient Preferences and a Clinical Tool for Evaluating for Sexual Function in Adolescent and Young Adult Survivors of Childhood Cancer
Brief Title: Sexual Function Screening in Childhood Cancer Survivors
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-1111.cc; P30CA046934 (NIH)
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Childhood Cancer; Survivorship; Sexual Dysfunction
MeSH Terms: conditions — Neoplasms; Sexual Dysfunction, Physiological | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- age 15-19: The investigators plan to complete 24 interviews with 12 in the age 15-19 cohort.The investigators will also ensure that at least 8 people from each sex are included in this study.
  Interventions: Other: Interviews
- age 20-24: The investigators plan to complete 24 interviews with 12 in the age 20-24 cohort. The investigators will also ensure that at least 8 people from each sex are included in this study.
  Interventions: Other: Interviews

INTERVENTIONS:
Other: Interviews — * Participation will serve as verbal consent.
  * Qualitative PRA will call participant to schedule either phone or in person interview. If via phone, the study PRA performing the interview, will remind them to find a private space to speak.
  * REDCap link will be sent for PROMIS SexFS Brief.
  * PRA will perform semistructured interview and guide Think-Aloud to complete the PROMIS SexFS Brief.
  * Participants will not submit responses to PROMIS SexFS Brief responses after completing the tool.

SUMMARY:
This is a qualitative research study involving semistructured interviews and Think-Aloud methodology during completion of a clinical screening tool. All participants will undergo the same semistructured interviews.

DETAILED DESCRIPTION:
The proposed research will explore patient-centered approaches to evaluating younger Adolescent/young adult Childhood cancer survivors for sexual dysfunction, including strategies for implementation and usability of thePatient-Reported Outcomes Measurement Information® v2.0 Brief Profile for Sexual Function and Satisfaction Brief, an existing adult screening tool. This study will include interviews with 24 patients age 15-24 who were diagnosed with cancer prior to age 18, and treated with chemotherapy, radiation and/or surgery and are now at least two years off therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to read and understand the postcard consent.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Age 15-24 at time of enrollment
4. History of cancer diagnosis, diagnosed at <18 years old
5. Off therapy (chemotherapy, surgery, radiation) for a minimum of 2 years
6. Sufficient cognitive functioning such that participants are able to complete study measures, as determined by their physician and research personnel.

Exclusion Criteria:

1. Developmental or intellectual disability, as determined by the patient's physician
2. Received neither chemotherapy nor radiation therapy
3. Non-English speaking
4. Non-English reading

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * Sample size
    * Max number of participants that can be enrolled is 30
    * Max number of participants that can be interviewed is 24
  * Gender Male and Female
  * Age Range 15-24
  * Demographic group English-speaking
  * General health status Pediatric cancer survivors (diagnosed at <18 years of age and now at least 2 years off therapy)
  * Geographic location Children's Hospital Colorado and University of Colorado Hospital
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Describe AYA CCS perspectives on implementation of screening for sexual dysfunction, including preferred modality, setting and timing for evaluating sexual dysfunction. | 1 year
  Qualitative interviews will be conducted by phone by a trained qualitative research interviewer. Interviews will be in-depth and semistructured, utilizing a combination of broad, open-ended questions and more specific probes. The interview guide was developed with the help of Dr. Michael Fisher, PhD, who has expertise in qualitative research methodology. The interviewer will take detailed field notes. This portion of the interview will last approximately 25-35 minutes and will be digitally recorded and professionally transcribed. After each interview, the interviewer will complete an Interview Summary Form, which will serve as a memoing tool and summarize initial themes or impressions that may be relevant to the research question.

SECONDARY OUTCOMES:
Assess AYA CCS perceptions of the PROMIS SexFS Brief, an existing adult clinical screening tool for sexual dysfunction, in a qualitative pilot study. | 1 year
  Participants will be asked to evaluate the PROMIS SexFS Brief, which will be emailed to them at the time of the interview via a unique/secure REDCap link. Participants will be given a choice of which version of the tool they complete (male or female). Participants will be asked to complete the PROMIS SexFS Brief via REDCap while completing Think-Aloud methodology. Via Think-Aloud, participants will be asked to verbalize their thoughts as they proceed through the task, which asks participants to verbalize their thoughts, without probing or additional explanations, as they undertake a task such as completing a clinical screening questionnaire. In accordance with recommendations for conducting Think-Aloud, participants will participate in a warm-up exercise unrelated to sexual dysfunction prior to completing Think-Aloud.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - Colorado School of Public Health, University of Colorado Denver, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No